CLINICAL TRIAL: NCT04350190
Title: A Prospective Multicenter Phase II Clinical Trial of Apatinib Mesylate Tablets Combined With PD-1 in the Treatment of Recurrent or Metastatic Nasopharyngeal Carcinoma
Brief Title: Apatinib Combined With PD-1 in the Treatment of Recurrent or Metastatic Nasopharyngeal Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Wei Jiang (Other)
Collaborators: Wuzhou Red Cross Hospital (Other); Guangxi Naxishan Hospital (Other); Laibin People's Hospital (Other); People's Hospital of Lingshan (Unknown)
Responsible Party: Sponsor-Investigator, Wei Jiang, Wei Jiang,MD,PhD, Guilin Medical University, China
Organization: Guilin Medical University, China (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GLMU-06
Record Dates: First submitted 2020-04-14; First posted 2020-04-16 (Actual); Last update posted 2023-01-13 (Actual); Status verified 2023-01

CONDITIONS: Nasopharyngeal Carcinoma
Keywords: Nasopharyngeal Carcinoma; Apatinib; PD-1; Second-line treatment; Overall response rate
MeSH Terms: conditions — Nasopharyngeal Carcinoma | interventions — apatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Apatinib combined with PD-1 (Experimental): Eligible patients begin to use apatinib mesylate tablets and PD-1, apatinib mesylate tablets at the recommended dose of 250mg,oral, QD, continuous administration, 4 weeks (28 days) as an observation cycle. Until the disease progressed or unbearable adverse reactions appeared. If missed medication occurs during the medication period, it is confirmed that the next medication time is less than 12 hours, then there will be no replenishment. The recommended dose of PD-1 is 200mg/time, Q2W, intravenous injection, 4 weeks (28 days) as an observation cycle, until disease progression or intolerable toxicity.
  Interventions: Drug: Apatinib mesylate tablet; Drug: PD-1

INTERVENTIONS:
Drug: Apatinib mesylate tablet — The dose of apatinib mesylate tablets is 250mg, oral, qd, continuous administration, 4 weeks (28 days) as an observation cycle.
Drug: PD-1 — The dose of PD - 1 is 200 mg/ time, intravenous injection, q2w, 4 weeks (28 days) for an observation period.

SUMMARY:
The study is to evaluate the clinical efficacy of apatinib mesylate tablets combined with PD-1 in the treatment of recurrent and metastatic nasopharyngeal carcinoma after IMRT with concurrent chemotherapy,including The Overall Response Rate (ORR), Progression-free survival (PFS),Overall survival (OS),and Toxicities.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

To determine the clinical efficacy of apatinib mesylate tablets combined with PD-1 in the treatment of recurrent and metastatic nasopharyngeal carcinoma.

SECONDARY OBJECTIVES:

Ⅰ.To explore the adjuvant medication regimen of recurrent and metastatic nasopharyngeal carcinoma.

Ⅱ.Provide high-level evidence-based medical evidence for the new individualized treatment strategy of nasopharyngeal carcinoma patients.

OUTLINE:

Eligible patients begin to use apatinib mesylate tablets and PD-1, apatinib mesylate tablets at the recommended dose of 250mg,orally, QD, continuous administration, 4 weeks (28 days) as an observation cycle. Until the disease progressed or unbearable adverse reactions appeared. If missed medication occurs during the medication period, it is confirmed that the next medication time is less than 12 hours, then there will be no replenishment. The recommended dose of PD-1 is 200mg/time, Q2W, intravenous injection, 4 weeks (28 days) as an observation cycle, until disease progression or intolerable toxicity.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients: 18-70 years old.
2. Pathologically diagnosed nasopharyngeal carcinoma.
3. Patients with nasopharyngeal carcinoma who have local recurrence after one comprehensive treatment (clinical examination found definite local residual: clear residual or cervical enlarged lymph node can be seen under electronic nasopharyngoscope).
4. Patients with nasopharyngeal carcinoma who have distant metastasis after one comprehensive treatment (found distant metastasis by liver ultrasound, chest X-ray, bone scan or other examination (such as CT, MRI or PET/CT) as the clinician considers appropriate.
5. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
6. Estimated survival ≥6 months.
7. The function of the main organs is good, that is, one week before joining the group, the following requirements are met:

   Blood routine examination:Hemoglobin > 80 g/L(no blood transfusion within 14 days);Neutrophils count > 1.5x10^9/L;Platelet count > 80x10^9/L; biochemical test:serum total bilirubin ≤1.5×ULN(upper limit of normal), ALT or AST≤3×ULN;Endogenous creatinine clearance ≥ 1.5×ULN;Acceptable clotting state: the international standardized ratio ((INR)), prothrombin time (PT) and activated partial thromboplastin time (APTT) of blood clots were less than 1.5 times of the upper limit of normal (ULN).
8. All women with fertility potential must undergo a urine or serum pregnancy test during screening and the results are negative.
9. The subjects voluntarily joined the study, signed the informed consent form, had good compliance and cooperated with the follow-up.

Exclusion Criteria:

1. Before treatment, MRI showed that the tumor may have invaded important blood vessels (such as enclosing the internal carotid artery / vein), or researchers have determined that the tumor is highly likely to invade important blood vessels and cause fatal massive bleeding during treatment.
2. There was a history of severe bleeding, and any bleeding events with a serious grade of 3 or more in CTCAE4.0 occurred within 4 weeks before screening.
3. Patients with hypertension who cannot be well controlled by antihypertensive therapy alone (systolic blood pressure > 140mmHg, diastolic blood pressure > 90mmHg); patients with a history of unstable angina pectoris; patients newly diagnosed with angina pectoris within 3 months or myocardial infarction within 6 months before screening; arrhythmias (including QTcF: ≥ 450ms in males, ≥ 470ms in females) require long-term use of antiarrhythmic drugs and New York Heart Association grade ≥ II cardiac insufficiency.
4. Positive urine protein.
5. Patients with abnormal blood coagulation and bleeding tendency (14 days before signing informed consent: INR is within the normal range without anticoagulant); patients treated with anticoagulants or vitamin K antagonists such as warfarin, heparin or their analogues; On the premise that the international standardized ratio of prothrombin time ((INR)) is less than 1.5, low-dose warfarin (1mg orally, once a day) or low-dose aspirin (daily dose not more than 100mg) is allowed for preventive purposes.
6. Arteriovenous thrombosis occurred within one year before screening, such as cerebrovascular accident (including temporary ischemic attack), deep venous thrombosis (except venous thrombosis caused by intravenous catheterization due to early chemotherapy) and pulmonary embolism.
7. Long-term unhealed wound or incomplete fracture.
8. Any factors that affect the oral drug, such as inability to swallow, chronic diarrhea and intestinal obstruction, etc.
9. For female subjects: women of childbearing age, it is not acceptable to use medically approved contraception during the study treatment period and within 6 months after the end of the study treatment period;Patients with positive serum or urine pregnancy test;Nursing patients.Male subjects: patients who did not undergo surgical sterilization or did not agree to use medically approved contraception during the study and within 6 months after the study.
10. Having a history of psychotropic substance abuse and unable to quit or having mental disorders.
11. Medical history of immunodeficiency, or other acquired, congenital immunodeficiency disease, or history of organ transplantation.Any symptomatic autoimmune disease (such as lupus, scleroderma, Crohn's disease, ulcerative colitis) that requires administration of >10mg of prednisone equivalent. Lower dose steroids for conditions such as hypophysitis are allowed.
12. Any serious harm to the subject's safety or evidence of significant medical illness that in the investigator's judgment will substantially increase the risk associated with the subject's participation in and completion of the study.
13. Any prior severe adverse event attributed to prior anti-PD1 therapy that, in the Principal investigator's opinion, would contraindicate pembrolizumab administration such as:Grade 2 or higher pneumonitis、Grade 4 AST or ALT elevation、Grade 3 or higher colitis; Known active infection with Hepatitis B Virus (HBV), Hepatitis C Virus (HCV), or HIV. Cleared HBV/HCV infection is not an exclusion, nor is HIV infection with cluster of differentiations 4 (CD4) counts >500 and an undetectable viral load.
14. Active bacterial, viral, or fungal infections, requiring systemic therapy apart from anti-viral maintenance therapy for HIV；or Uncontrolled activity infected.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2021-01-14 (Actual); Primary Completion 2022-09-15 (Actual); Study Completion 2022-09-15 (Actual)

PRIMARY OUTCOMES:
Overall Response Rate (ORR) | Up to 24 months
  To evaluate ORR every 6-8 weeks after initiation of treatment.

SECONDARY OUTCOMES:
Progression-free survival (PFS) | Up to 24 months
  The time from the first day of therapy to locoregional relapse, distant relapse or tumor-related death
Overall survival (OS) | Up to 24 months
  The time from the first day of therapy to death or last follow-up
Number of Participants with Adverse Events | Up to 24 months
  Incidence of acute and late toxicity

CONTACTS AND LOCATIONS:
Overall Officials: Wei Jiang, Ph.D., Study Director — Guilin Medical University, China
Locations (5):
- China (5):
  - Guilin Medical University, Guilin, Guangxi
  - Nanxishan Hospital of Guangxi Zhuang Autonomous Region, Guilin, Guangxi
  - People's Hospital of Laibin, Laibin, Guangxi
  - People's Hospital of Lingshan, Linshan, Guangxi
  - Wuzhou Red Cross Hospital, Wuzhou, Guangxi

REFERENCES:
- [Derived] Mo Y, Pan Y, Zhang B, Zhang J, Su Y, Liu Z, Luo M, Qin G, Kong X, Zhang R, Pan Y, Liang Y, Wang D, Wei Y, Chen H, Jiang W. Apatinib combined with camrelizumab in the treatment of recurrent/metastatic nasopharyngeal carcinoma: a prospective multicenter phase II study. Front Immunol. 2024 Jan 3;14:1298418. doi: 10.3389/fimmu.2023.1298418. eCollection 2023. PMID 38239359